CLINICAL TRIAL: NCT00884767
Title: Characterization and Research of Predictive Markers of Neurotoxicity During Treatment With Oxaliplatin in Colorectal Carcinoma: a Genetic and Proteomic Approach. Phase II Multicenter Study
Brief Title: Biomarkers in Predicting Neurotoxicity in Patients With Colorectal Cancer Receiving Oxaliplatin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000633477; CPP-NEUROTOXALI; CPP-CPP340; INCA-RECF0453; EUDRACT-2007-001287-75
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Chemotherapeutic Agent Toxicity; Colorectal Cancer; Neurotoxicity
Keywords: neurotoxicity; chemotherapeutic agent toxicity; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neurotoxicity Syndromes; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Gene Expression Profiling; Pharmacogenomic Testing

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Genetic: gene expression analysis
Genetic: protein expression analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis
Other: pharmacogenomic studies

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving oxaliplatin for cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to neurotoxicity.

PURPOSE: This phase II trial is studying biomarkers in predicting neurotoxicity in patients with colorectal cancer receiving oxaliplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate predictive genetic, proteomic, and/or neurotrophic markers with neurological manifestations related to the administration of oxaliplatin in patients with colorectal carcinoma.

Secondary

* Differentiate between risk factors predictive of acute and chronic neurotoxicity.
* Establish a possible relationship between acute and chronic neurotoxicity.

OUTLINE: This is a multicenter study.

Patients receive oxaliplatin every 2 weeks as part of a FOLFOX chemotherapy regimen.

Blood samples are collected 15 days prior to beginning chemotherapy, prior to each course of chemotherapy, and at 1 month after completion of chemotherapy for pharmacogenetic and laboratory biological studies. Patients with chronic neurotoxicity undergo additional blood sample collection at 3, 6, 9, and 12 months after completion of chemotherapy. Samples are analyzed for the detection of gene variants involved in the oxalate and fluorouracil metabolic pathway; neurotrophic factors; proteomic analysis of plasma proteins and peptides; and for biological testing of neurotoxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer
* Requires treatment with oxaliplatin (as part of a FOLFOX regimen)
* No brain metastases or symptomatic meningitis

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 3 months
* ANC ≥ 1 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* Transaminases ≤ 3 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior or concurrent clinical neuropathy (regardless of the etiology)
* No dihydropyrimidine dehydrogenase deficiency
* No psychiatric illness that would preclude comprehension of the study or of the informed consent
* No other severe illness that may worsen during treatment, including unstable cardiac disease, myocardial infarction within the past 6 months, or active uncontrolled infection
* No psychological, social, familial, or geographical reason that would preclude study follow-up
* Other cancer within the past 5 years allowed provided treatment did not include platinum derivatives or taxanes

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior chemotherapy allowed (except for platinum derivatives or taxanes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Correlation of genetic profiles and peptide, protein, and neurotrophic factors with neurological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Erick Gamelin, MD, Principal Investigator — Institut Cancerologie de l'Ouest
Locations (1):
- Centre Paul Papin, Angers, France